CLINICAL TRIAL: NCT04448691
Title: "SIMULATION MODELING OF CORONARY ARTERY DISEASE: A TOOL FOR CLINICAL DECISION SUPPORT"
Acronym: SMARTool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Collaborators: University of Zurich (Other); Turku University Hospital (Other Government); Azienda USL 12 Versilia (Other); Federico II University (Other); Institut Catala de Salut (Other Government); National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Silvia Rocchiccioli, Project Coordinator, Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23534
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Management/Treatment of Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: prospective study with serial CCTA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCTA (Other): Suspected coronary disease patients enrolled in EVINCI trial with CCTA where recalled for follow up CCTA and blood sampling
  Interventions: Diagnostic Test: CCTA

INTERVENTIONS:
Diagnostic Test: CCTA — requested follow up CCTA

SUMMARY:
Coronary atherosclerosis (ATS) is a degenerative-inflammatory artery pathology underlying the different clinical manifestations of coronary heart disease (CHD), from stable angina due to constrictive plaque growth obstructing artery lumen, to acute coronary syndrome (ACS), secondary to abrupt lumen occlusion by atherothrombosis at the site of a ruptured or eroded plaque.

Major coronary adverse events (MACE) are known to be related to local factors, the so called "high risk plaque" characterized by large lipid-necrotic core with a thin fibrous cap, intraplaque hemorrhage, rupture, erosion, and to systemic, patient-specific, factors, contributing to the atherogenic genotype/phenotype of the so called "high risk patient", presenting with an abnormally activated thrombogenic and/or inflammatory state or increased plasma levels of atherogenic lipid species.

The huge social and economic impact of CHD in western and developing countries is primarily due to the difficulty to identify and predict, in the clinical context, which "high risk plaque" in which "high risk patient" will cause, independently of stenosis severity, an acute coronary event such as myocardial infarction or sudden coronary death, which are often the first manifestations of CHD in a large proportion of otherwise asymptomatic subjects. Plaque burden, compared to stenosis, is recognized as a better predictor of ACS and coronary CT angiography (CCTA) is considered as the optimal non-invasive coronary imaging modality to assess and quantify plaque burden and to evaluate the functional significance of a stenosis, by computationally estimating fractional flow reserve. Moreover, molecular studies of CHD patients have mostly examined associations with clinical cardiovascular outcomes: associations with coronary ATS assessed by quantitative CCTA may provide insight into the pathophysiological role of several molecular species in plaque formation and growth, and elucidate their potential role as discriminative biomarkers of CHD.

Based on these considerations, aim of this study is to collect and analyze all patient-specific clinical and epidemiological data and patient phenotype and genotype blood-derived molecular information, and to combine them with local high resolution non-invasive CCTA imaging of actual plaque burden as well as, prospectively, of its increase or de novo formation over a clinically relevant timespan. The expected result, following local and systemic data integration and modeling, is to optimize early diagnosis and risk stratification of CHD beyond current clinical models and scores and to help improving primary and secondary prevention of MACE. The overall design of this diagnostic and prognostic framework has been proposed to Horizon 2020 EU Call PHC30 and approved by the European Commission (Grant Agreement PHC30-689068). The Consortium includes major clinical European University Hospitals specialized in CHD imaging and treatment and the project study has obtained the endorsement of the European Society of Cardiovascular Imaging.

ELIGIBILITY:
Inclusion Criteria:

1. male and female subjects
2. aged 45-75 years
3. caucasian population
4. submitted to CCTA for suspected CHD between 2009 and 2012 (in the context of EVINCI and ARTreat FPVII studies) at the Hospitals reported in "SMARTool Clinical Center" document and satisfying the elegibility criteria reported above
5. submitted to clinical Follow-up in the last 6 months with stable clinical conditions and documented CHD or persistent intermediate/high probability of CHD
6. Signed informed consents (clinical and genetic)

Exclusion Criteria:

1. Multi-vessel severe disease (3 vessels and/or LM disease with >90% stenosis).
2. Severe coronary calcification (CAC score > 600).
3. Having undergone surgical procedures related to heart diseases (CABG, valve replacement, CRT or CRTD treatment, any surgery of the heart or arteries).
4. Documented MACE at history (myocardial infarction, severe heart failure, recurrent angina) in the last 6 months with/without revascularization
5. Documented severe peripheral vascular disease (carotid, femoral)
6. Surgery of carotid and/or peripheral arteries or cerebral ischemic attack
7. History/surgery of Abdominal Aortic Aneurysm(AAA).
8. Severe Heart failure (NYHA Class III-IV)
9. LV dysfunction (left ventricle EF <40%).
10. Atrial fibrillation.
11. Lack of written informed consent (clinical consent and/or genetic consent)
12. Pregnancy (evaluated by urine test) and breastfeeding
13. Active Cancer
14. Asthma
15. Severe untreated Hypertension (arterial blood pressure ≥ 170/110 mmHg)
16. Cardiomyopathy or congenital heart disease
17. Significant valvular disease (hemodynamically significant valvular stenosis or insufficiency by echoDoppler)
18. Renal dysfunction (creatinine > 1.3 mg/dL)
19. Chronic Kidney Disease (eGFR < 30 ml/min/1.73 m2)
20. Hepatic failure (at least 3 of the following: albumin < 3.5 g/dL; prolonged prothrombin time-PT; jaundice; ascites)
21. Waldenstrom disease
22. Multiple myeloma
23. Autoimmune/Acute inflammatory disease
24. Previous severe adverse reaction to iodine contrast agent
25. Positivity at blood tests for HIV, Hepatitis B and C (CRF number 1-clinical evaluation)

    -

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
coronary artery disease progression assessed by CCTA | 6 years CCTA follow up

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caselli C, De Caterina R, Smit JM, Campolo J, El Mahdiui M, Ragusa R, Clemente A, Sampietro T, Clerico A, Liga R, Pelosi G, Rocchiccioli S, Parodi O, Scholte A, Knuuti J, Neglia D; EVINCI and SMARTool. Triglycerides and low HDL cholesterol predict coronary heart disease risk in patients with stable angina. Sci Rep. 2021 Oct 20;11(1):20714. doi: 10.1038/s41598-021-00020-3. PMID 34671067
- [Derived] El Mahdiui M, Smit JM, van Rosendael AR, Neglia D, Knuuti J, Saraste A, Buechel RR, Teresinska A, Pizzi MN, Roque A, Magnacca M, Mertens BJ, Caselli C, Rocchiccioli S, Parodi O, Pelosi G, Scholte AJ. Sex differences in coronary plaque changes assessed by serial computed tomography angiography. Int J Cardiovasc Imaging. 2021 Jul;37(7):2311-2321. doi: 10.1007/s10554-021-02204-4. Epub 2021 Mar 10. PMID 33694122
- [Derived] Sbrana S, Campolo J, Clemente A, Bastiani L, Cecchettini A, Ceccherini E, Caselli C, Neglia D, Parodi O, Chiappino D, Smit JM, Scholte AJ, Pelosi G, Rocchiccioli S. Blood Monocyte Phenotype Fingerprint of Stable Coronary Artery Disease: A Cross-Sectional Substudy of SMARTool Clinical Trial. Biomed Res Int. 2020 Jul 27;2020:8748934. doi: 10.1155/2020/8748934. eCollection 2020. PMID 32802883
- See also: H2020 project website — http://www.smartool.eu